CLINICAL TRIAL: NCT06919237
Title: Chronic Adaptations in Cardiovagal Modulation and Cardiorespiratory Fitness in Patients With Coronary Artery Disease to a 12-week Heart Rate Variability-guided Training vs Traditional Aerobic Prescription Program: Study Protocol for a Randomized Controlled Trial
Brief Title: Effects of Heart Rate Variability-guided Training vs Standard Aerobic Prescription on Cardiovagal Modulation and Cardiorespiratory Fitness in Coronary Artery Disease
Acronym: ParaDox
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Faculdade de Motricidade Humana (Other)
Collaborators: Fundação para a Ciência e a Tecnologia (FCT) (Unknown)
Responsible Party: Principal Investigator, Manuel Pedro, Principal Investigator (PhD project), Faculdade de Motricidade Humana
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ParaDox
Record Dates: First submitted 2025-03-30; First posted 2025-04-09 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-03

CONDITIONS: Coronary Arterial Disease (CAD)
Keywords: Exercise prescription; arterial stiffness; heart rate variability; autonomic activity; maximal oxygen consumption; moderate-intensity continuous training; high-intensity interval training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- HIIT (training/Behavioral) (Experimental): Over the first 4 weeks, participants will perform 4 bouts of 2 min of high-intensity exercise at 80-90% heart rate reserve (HRR), during the next 4 weeks, participants will perform 6 bouts of 2 min of high-intensity exercise at 80-90%HRR, while in the last 4 weeks participants will perform 6 bouts of 2 min of high-intensity exercise at 90%HRR). Exercise bouts will be interspersed by 2 min of active recovery at 50-60% HRR.
  Interventions: Other: HIIT Intervention
- MICT (training/Behavioral) (Experimental): Over the first 4 weeks participants in MICT will perform continuous exercise at 50-60% HRR (2x10'), during the next 4 weeks participants will perform continuous exercise at 50-60% HRR (2x12'), while in the last 4 weeks participants will perform continuous exercise at 60-70% HRR (2x15').
  Interventions: Other: MICT Intervention
- HRV-Guided Training (training/Behavioral) (Experimental): Following a 10-day initial characterization period, where the HRV is measured with plethysmography continually during the night, with "Whoop" (https://www.whoop.com) device, the individual HRV profile is defined, still, participants will use the Whoop during all intervention to allow the updating of HRV profile. Then, considering the daily individual autonomic regulation, following a decision-making schema modiﬁed from Kiviniemi et al., (2007) [21], exercise intensity will be defined for the training session, i.e., if LnRMSSD7day-roll-avg remained inside the smallest worthwhile change (SWC) (SWC = 0.5 × standard deviation), high intensity or moderate-intensity training sessions is prescribed, if LnRMSSD7day-roll-avg fell outside SWC, low intensity or rest is prescribed, leading to different workloads from the predefined training programs.
  Interventions: Other: HRV-Guided Intervention

INTERVENTIONS:
Other: HIIT Intervention — Over the first 4 weeks, participants will perform 4 bouts of 2 min of high-intensity exercise at 80-90% heart rate reserve (HRR), during the next 4 weeks, participants will perform 6 bouts of 2 min of high-intensity exercise at 80-90%HRR, while in the last 4 weeks participants will perform 6 bouts of 2 min of high-intensity exercise at 90%HRR). Exercise bouts will be interspersed by 2 min of active recovery at 50-60% HRR.
  Arms: HIIT (training/Behavioral)
Other: MICT Intervention — Over the first 4 weeks participants in MICT will perform continuous exercise at 50-60% HRR (2x10'), during the next 4 weeks participants will perform continuous exercise at 50-60% HRR (2x12'), while in the last 4 weeks participants will perform continuous exercise at 60-70% HRR (2x15').
  Arms: MICT (training/Behavioral)
Other: HRV-Guided Intervention — Following a 10-day initial characterization period, where the HRV is measured with plethysmography continually during the night, with "Whoop" (https://www.whoop.com) device, the individual HRV profile is defined, still, participants will use the Whoop during all intervention to allow the updating of HRV profile. Then, considering the daily individual autonomic regulation, following a decision-making schema modiﬁed from Kiviniemi et al., (2007) [21], exercise intensity will be defined for the training session, i.e., if LnRMSSD7day-roll-avg remained inside the smallest worthwhile change (SWC) (SWC = 0.5 × standard deviation), high intensity or moderate-intensity training sessions is prescribed, if LnRMSSD7day-roll-avg fell outside SWC, low intensity or rest is prescribed, leading to different workloads from the predefined training programs.
  Arms: HRV-Guided Training (training/Behavioral)

SUMMARY:
Coronary artery disease (CAD) is associated with autonomic dysfunction and is characterized by reduced heart rate variability (HRV) and impaired heart rate recovery. Regular exercise improves cardiovascular outcomes in CAD, with high-intensity interval training (HIIT) showing superior benefits compared to moderate-intensity continuous training (MICT). However, the full potential of exercise is not used in the clinical context since some of the training principles are neglected, contributing to a high number of exercise non-responders. HRV-guided training has been identified as an alternative prescription technique for cardiovascular endurance exercise and has contributed to greater improvements compared to standard prescriptions. Thus, this study aims to assess the chronic effects of exercise on cardiovagal modulation, baroreflex sensitivity, arterial stiffness, and cardiorespiratory fitness in patients with CAD, specifically determining whether heart rate variability-guided training yields different outcomes compared to a traditional prescription in a 12-week exercise intervention.

A total of 48 participants, will be recruited and randomized into one of 3 groups: high-intensity interval training (HIIT), moderate-intensity continuous training (MICT), and HRV-guided training. The intervention will consist of 12 weeks of supervised exercise, with 3 weekly sessions. Participants in the HRV-guided training group will have their exercise intensity adjusted based on their individual HRV profiles. Moderate- or high-intensity sessions are prescribed when the 7-day rolling average of LnRMSSD remains within the smallest worthwhile change (SWC). If it falls outside the SWC, low-intensity sessions or rest are recommended. In the HIIT group, sessions will consist of 4 bouts of 2 minutes at 80-90% HRR during the first 4 weeks, increasing to 6 bouts of 2 minutes at the same intensity in weeks 5-8, and progressing to 6 bouts of 2 minutes at 90% HRR in the final 4 weeks. In the MICT group, participants will perform continuous sessions starting with 2x10 minutes at 50-60% HRR in the first 4 weeks, progressing to 2x12 minutes at the same intensity in weeks 5-8, and increasing to 2x15 minutes at 60-70% HRR in the final phase. Cardiovagal modulation, cardiorespiratory fitness, BRS, and AS will be assessed at the baseline and after the 12 weeks of intervention.

Most cardiac rehabilitation programs use the "one-size-fits-all" approach, which is a limitation of the literature, leading to a large number of exercise nonresponders to changes in cardiorespiratory fitness. HRV-guided training seems to be a more individualized method of aerobic prescription and may lead to greater improvements in cardiorespiratory fitness and in cardiovagal modulation. This study will contribute to generate evidence regarding aerobic exercise prescription in cardiac rehabilitation.

DETAILED DESCRIPTION:
Background

Coronary artery disease (CAD) is characterized by the inability to adequately supply blood and oxygen to the heart, often resulting from the formation of atherosclerotic plaques within the arterial lumen. This inflammatory, multifactorial condition can impair the autonomic nervous system (ANS), disrupting the balance between the sympathetic and parasympathetic pathways and leading to autonomic dysfunction. Key indicators of this dysfunction include reduced heart rate variability (HRV) and delayed heart rate recovery, both of which signify heightened sympathetic activity and diminished parasympathetic activity. These changes predict worse cardiovascular outcomes in CAD patients, as the ANS compensates for myocardial ischemia and hypoxia by increasing sympathetic drive and reducing vagal activity to preserve cardiac contractility and output. This imbalance triggers a cascade of neurohumoral alterations affecting the cardiovascular, peripheral vascular, and renal systems, further exacerbating disease progression.

Regular exercise is known to play an important role in the prevention, management, and treatment of CAD, mainly through the preservation of endothelial function but also through the improvement of cardiovagal modulation and neurocardiovascular stress reactivity and by the increase in cardiorespiratory fitness. Patients with stable CAD should undergo a cardiac rehabilitation program to fulfill exercise guidelines. Protocols may vary in mode, intensity, frequency, and duration, whereas the most recommended types of exercise are walking and cycling, with intensities between 40-80% of VO2peak associated with increases in exercise capacity by 11-36%. Recent studies demonstrated that high-intensity interval training (HIIT) compared with moderate-intensity continuous training (MICT) promotes higher adaptation in VO2max and in post-exercise heart rate recovery, HIIT has also demonstrated to contribute to the restoration of endothelial function and autonomic balance, inducing reverse cardiac remodeling and increasing left ventricle morphology and function. However, MICT demonstrates higher adherence because it is a safer and more effective approach. Nevertheless, despite the known non-pharmacological benefits of exercise, recent studies demonstrate that more than 15% of the patients with CAD are exercise non-responders to increases in VO2max , i.e., an increase of 3.5 ml/kg/min in VO2max, which has been associated with a 10% decrease in all-cause of mortality and cardiovascular mortality, however the greater the increases in VO2max the greater the reduction in the risk.

Exercise individualization is increasing among apparently healthy populations due to the ease of the use of cellphone applications. Recently, HRV-guided training has been identified as an alternative prescription technique for cardiovascular endurance exercise prescription, this prescription technique demonstrated to contribute to greater improvements in endurance athletes. HRV-guided training concerns to exercise prescribed based on daily changes in HRV, depending on thresholds constructed at the individual level. After an initial characterization period, where the HRV after waking up is measured, the individual HRV profile is defined. Then, considering the resting values of HRV, exercise intensity will be determined for the training session, i.e., if LnRMSSD7day-roll-avg remained inside the smallest worthwhile change (SWC) (+), high-intensity or moderate-intensity training sessions is prescribed, and if LnRMSSD7day-roll-avg fell outside SWC (-), low intensity or rest is prescribed. This prescription technique leads to different workloads from the predefined training programs.

To the best of our knowledge, no study has yet compared the chronic effects of two different exercise protocols on cardiovagal modulation, and cardiorespiratory fitness in patients with CAD. Thus, this research aims to compare the chronic adaptations on cardiorespiratory fitness, cardiovagal modulation, baroreflex sensitivity (BRS), and arterial stiffness (AS) of two different techniques of exercise prescription (traditional vs individualized) and two training methods (HIIT vs MICT) in patients with CAD. We hypothesize that exercise individualization will promote higher adaptations in cardiovagal modulation, cardiorespiratory fitness, BRS and AS in patients with CAD, compared with traditional prescription.

Methods

Study design This longitudinal randomized trial will consist of comparing the effects of different exercise prescription techniques and different methods of exercise prescription (traditional MICT, traditional HIIT, and HRV-guided training) would exhibit differences in chronic adaptations in cardiorespiratory fitness, cardiovagal modulation, and BRS in patients with CAD. The study will consist of 12 weeks of supervised exercise with 3 sessions per week. This study protocol was submitted to the Faculty of Human Kinetics Institutional Review Board.

Sample size

Assuming a change in VO2max of 3.5 mL/kg/min to be clinically relevant, α = 0.05, 1-β = 0.80, an expected dropout of 15% for 12 weeks, and a chosen medium effect size of 0.25 due to gaps in the literature, the calculations yielded a total minimum of 48 participants (16 per group) (G*Power, version 3.1.9.4), however, the sample size will be updated, if necessary, after a pilot study consisting of 12 participants, 4 per group, (48x0.25=12).

Recruitment

Recruitment will be performed mainly at the Coronary Club of Lisbon (CORLIS) (phase III) at the Faculty of Human Kinetics and at the Hospital of Santa Cruz in Lisbon.

Measurements

All study measurements will be collected at the Faculty of Human Kinetics, University of Lisbon. Assessments of cardiopulmonary exercise test (CPET), cardiovagal modulation, body composition, and arterial stiffness, will be conducted both at baseline and after the 12-week intervention period. Participants will be requested to be fasted (> 4h), abstain from foods/drinks containing caffeine and alcohol (> 12h), and refrain from strenuous exercise (> 24h) before assessments, post-intervention assessments will be scheduled for the same time that baseline. The measures will follow the following order body composition, cardiovagal modulation (and baroreflex sensitivity), local and regional arterial stiffness, cardiopulmonary test, and post-maximal exercise cardiovagal modulation (and baroreflex sensitivity), and local and regional arterial stiffness.

Randomization

Baseline evaluation will be done before randomization, thus neither participants nor fieldwork staff will know the group assignment at this point. Due to the nature of the intervention, it will not be possible to blind participants after baseline assessments. After the baseline assessments, block randomization by group with balanced blocks of 12 participants will be performed by a researcher not involved in recruitment or data collection using REDCap (https://imm.medicina.ulisboa.pt/group/redcap/redcap_v7.6.7/). The participants will be randomly allocated to one of the three groups: HIIT, MICT, and HRV-guided training.

Exercise intervention

Exercise intervention will have a 12-week duration, with 3 sessions per week on non-consecutive days for all 3 groups and will be carried out at the Faculdade de Motricidade Humana. Certified exercise physiologists will supervise sessions. Heart rate will be monitored during all sessions with an HR monitor (S810i Polar, Polar Electro, Kempele, Finland; sampling rate 1000 Hz). All sessions will include a 10-minute warm-up, an aerobic component, a strength component, and a cool-down for both groups. The warm-up will focus on increasing HR, improving mobility, and performing preparatory stretches for the conditioning component. The strength component will consist of 6 arm and 2 leg machines with 2 sets of 8 to 12 reps at 50-60% 1RM per machine. The cool-down will transition from the conditioning component to the stretching phase, consisting of static and dynamic stretching exercises for all major muscle groups. Warm-up, strength component and coold-down will be standardized for the 3 groups. Sessions will be deemed completed when at least 83.3% (30 out of 36 sessions i.e. minimum adherence = 83.3%) of the prescribed exercise sessions have been successfully performed (reached the programmed intensity). The aerobic component in all groups will follow linear periodization. Volume and/or intensity will increase every 4 weeks.

Data analysis

All HRV analyses will be performed offline using the FisioSinal software built-in Matlab [25]. Time-domain and spectral power analyses will be conducted using 2-min time bins. Ectopic heartbeats (M = 1, SD = 4 b.min-1) will be excluded from the final analysis. The time-domain statistics used to characterize HRV will be SDNN and RMSSD. Non-linear time-domain parameters will be derived from the Poincaré plot including SD1 and SD2. The time-frequency domain analysis will be conducted using the Daubechy-12 discrete wavelet algorithm. Wavelet analysis will be chosen instead of fast Fourier transform as it is better suited to characterize the acute responses of the autonomic nervous system during exercise. The baroreflex effectiveness index (BEI) and BRS will be estimated using the spontaneous sequence method. Briefly, the method casts about adjacent oscillations (ramps) in systolic blood pressure (SBP; > 1 mmHg) and RR and ( > 4 ms). BRS will be defined as the average of the BRS slopes. BEI will be calculated as the total number of BRS events divided by the total number of BP ramps observed during the 2-minute time-bin.

Statistical methods

Statistical tests will be performed in R (R studio Version 4.2.2). Descriptive statistics will be employed to analyze demographic and clinical variables measured at the baseline for each group. Categorical variables will be presented using frequencies and percentages, while continuous variables will be expressed as mean ± standard deviation (or median and range).

For the primary and secondary outcomes, data will undergo analysis using linear mixed models in R, and lme4. The fixed effects will be defined as the moment of intervention, and group, and the random intercept will be defined as each participant. Parameter estimation will utilize restricted maximal likelihood and the Kenward-Roger approximation for degrees of freedom will be applied for evaluating significance, ensuring optimal type I error rates. Secondary analyses will explore adjustments for protocol deviations through a per-protocol analysis. Post a significant interaction, pairwise comparisons will be conducted with a Bonferroni adjustment. For main and interaction effects, partial eta squared (η2) will be computed as an effect size estimate. Effect sizes for pairwise comparisons will be reported as Cohen's d, complemented by 95% confidence intervals for mean differences. All statistical analyses will be conducted using R software, with a significant level of α = 0.05.

ELIGIBILITY:
Inclusion Criteria:

* aged over 18 years;
* had angiographically documented CAD in at least one major epicardial vessel;
* clinical evidence of CAD in the form of previous myocardial infarction;
* clinical evidence of CAD in the form of coronary revascularization (coronary artery bypass grafting or percutaneous coronary intervention);
* clinical evidence of CAD in the form of angina pectoris.

Exclusion Criteria:

* heart failure;
* cardiac implantable defibrillators;
* resynchronizing devices;
* inability to comply with guidelines for participation in exercise testing and training.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Cardiovagal modulation | pre and post intervention (12 weeks) assessments
  The R-R intervals will be derived from beat-to-beat blood pressure pulse intervals using finger plethysmography (Finapres Nova, Amsterdam, Netherlands), during all measures. Finger plethysmography-derived peak-to-peak intervals are highly correlated with electrocardiogram R-R intervals, with similar variability. The upstroke is determined using the pressure signal with a resolution of 2 ms, and the interval between the two consecutive upstrokes is measured. In the frequency domain, the two primary components are low-frequency (LF: 0.04-0.15 Hz) and high-frequency (HF: 0.15-0.40 Hz) spectra. Heart rate variability measures provide information primarily on vagal modulation with the LF power spectrum reflecting both sympathetic and parasympathetic modulation and HF reflecting the parasympathetic modulation of the R-R intervals. The LF/HF ratio is used as an indicator of sympathovagal dominance.
Cardiorespiratory fitness | pre and post intervention (12 weeks) assessments
  An incremental CPET will be performed on a treadmill (Pulsar 3p, HP Cosmos) with mixing-chamber gas exchange measurements (Quark RMR w/CPET, Italy), according to Bruce modified protocol. A 12-lead electrocardiogram will be continuously monitored, and blood pressure will be assessed by auscultation using an aneroid sphygmomanometer. A cardiologist and an exercise physiologist will supervise the CPET.
  Before each test, the gas analyzer will be calibrated using ambient air standard calibration gases of known concentrations (16,7% O2 and 5,7% CO2). The turbine flowmeter of Cosmed will be calibrated with a 3L syringe. Data will be analyzed in 20 s average, and peak VO2 will be defined as the highest value attained in the last minute of effort

SECONDARY OUTCOMES:
Baroreflex sensitivity | pre and post intervention (12 weeks) assessments
  Spontaneous sequence method will be used to estimate BRS through the baroreflex module of FisioSinal [25]. This method emits about adjacent oscillations (ramps) in R-R and ( > 4 ms) and systolic blood pressure (SBP) (SBP; > 1 mmHg). Beat-to-beat SBP will be recorded using finger plethysmography (Finapres Measurement Systems, Amsterdam, Netherlands). A BRS event was defined as the overlap of BP ramps with concordant changes in R-R intervals. Hence, BRS will be defined as the average of the BRS slopes.
Local arterial stiffness | pre and post intervention (12 weeks) assessments
  Carotid arterial stiffness indices will be assessed using eTRACKING technology (Arietta V60, Hitachi Aloka Medical Ltd, Mitaka-shi, Tokyo, Japan), using a 7.5 MHz linear array probe incorporating a 5 MHz Doppler transducer. In longitudinal view, the probe will be manipulated so that the intima of the artery is imaged clearly from both the anterior and posterior walls and a single scan line is aligned perpendicularly to the vessel walls at a site 20 mm proximal to the carotid bulb. On-screen cursors will be placed on the anterior and posterior intima-media borders to enable tracking of both walls. The corresponding displacement waveforms and diameter curve will be calculated using high-resolution online wall tracking ("E-track" technology), with a sampling rate of 1 kHz. Arterial pressure waveforms were obtained automatically in real-time by calibrating peak and bottom values with SBP and DBP measured with sphygmomanometry, as previously validated.
Regional Arterial Stiffness | pre and post intervention (12 weeks) assessments
  Carotid femoral PWV, carotid-radial PWV, and femoral dorsalis PWV will be measured using a non-invasive automatic device (Complior, Alam Medical, France) with participants lied supine on a cushioned table. The common carotid artery, femoral, radial and dorsalis artery pressure waveforms will be recorded using 4 piezoelectric pressure mechanotransducers placed on each artery. The travel time distance will be defined as the tape measured distance over the body surface between the 2 recording sites of interest with distance being corrected by 0.8 factor for carotid femoral. All measurements will be performed by the same operator on the right side of the body after 10 pulse waveforms of enough quality (> 90%).

OTHER OUTCOMES:
Body composition | pre and post intervention (12 weeks) assessments
  Dual-energy X-ray absorptiometry (DXA) (Hologic Explorer-W, fan-beam densitometer, software QDR for Windows version 12.4, Waltham, USA) will be used to estimate total and regional fat mass, lean body mass, bone mineral content, and density. A whole-body scan will be performed, and the attenuation of X-rays pulsed between 70 and 140 kV synchronously with the line frequency for each pixel of the scanned image that will be measured. Abdominal and gynoid body fat mass will be measured through partial analyses of the DXA scan, based on regions of interest set by default in the DXA settings.
Free living physical activity | during one week
  ActiGraph GT9X accelerometers will be used to track daily physical activity (ActiGraph, Pensacola, FL). Participants will be required to wear the accelerometer on their non-dominant wrist to control their level of physical activity. During the intervention phase, participants will be asked to maintain their usual patterns of physical activity. Actilife®software (v.6.9.1; Fort Walton Beach, FL) will be used for device activation and download, while an open-source R package called GGIR version 2.6 will be used for processing. The accelerometer data will yield measures of time spent in sedentary behavior, volume, and intensity of physical activity (total minutes at light, moderate, and vigorous intensity, total counts, and counts/minute), and how each of these behaviors is compounded (i.e., periods spent engaging in physical activity or sedentary behavior).

CONTACTS AND LOCATIONS:
Overall Officials: Helena Santa-Clara, PhD, Principal Investigator — Faculdade de Motricidade Humana
Locations (1):
- Faculdade de Motricidade Humana, Lisbon, Lisbon District, Portugal

REFERENCES:
- [Background] Carrasco-Poyatos M, Gonzalez-Quilez A, Altini M, Granero-Gallegos A. Heart rate variability-guided training in professional runners: Effects on performance and vagal modulation. Physiol Behav. 2022 Feb 1;244:113654. doi: 10.1016/j.physbeh.2021.113654. Epub 2021 Nov 20. PMID 34813821
- [Background] Khan H, Kunutsor S, Rauramaa R, Savonen K, Kalogeropoulos AP, Georgiopoulou VV, Butler J, Laukkanen JA. Cardiorespiratory fitness and risk of heart failure: a population-based follow-up study. Eur J Heart Fail. 2014 Feb;16(2):180-8. doi: 10.1111/ejhf.37. Epub 2013 Dec 14. PMID 24464981
- [Background] Kang SJ, Ko KJ. Association between resting heart rate, VO2max and carotid intima-media thickness in middle-aged men. Int J Cardiol Heart Vasc. 2019 Mar 29;23:100347. doi: 10.1016/j.ijcha.2019.100347. eCollection 2019 Jun. PMID 30976652
- [Background] Epelde F. Current Status, Challenges, and Future Directions in Cardiac Rehabilitation. Medicina (Kaunas). 2024 Feb 25;60(3):388. doi: 10.3390/medicina60030388. PMID 38541114
- [Background] Ribeiro PAB, Boidin M, Juneau M, Nigam A, Gayda M. High-intensity interval training in patients with coronary heart disease: Prescription models and perspectives. Ann Phys Rehabil Med. 2017 Jan;60(1):50-57. doi: 10.1016/j.rehab.2016.04.004. Epub 2016 Jun 23. PMID 27346629
- [Background] Pinto R, Angarten V, Santos V, Melo X, Santa-Clara H. The effect of an expanded long-term periodization exercise training on physical fitness in patients with coronary artery disease: study protocol for a randomized controlled trial. Trials. 2019 Apr 11;20(1):208. doi: 10.1186/s13063-019-3292-9. PMID 30975195
- [Background] Mattioni Maturana F, Soares RN, Murias JM, Schellhorn P, Erz G, Burgstahler C, Widmann M, Munz B, Thiel A, Niess AM. Responders and non-responders to aerobic exercise training: beyond the evaluation of V O2max. Physiol Rep. 2021 Aug;9(16):e14951. doi: 10.14814/phy2.14951. PMID 34409753
- [Background] Santa-Clara H, Fernhall B, Mendes M, Sardinha LB. Effect of a 1 year combined aerobic- and weight-training exercise programme on aerobic capacity and ventilatory threshold in patients suffering from coronary artery disease. Eur J Appl Physiol. 2002 Oct;87(6):568-75. doi: 10.1007/s00421-002-0675-4. Epub 2002 Jul 30. PMID 12355198
- [Background] Rakebrandt F, Palombo C, Swampillai J, Schon F, Donald A, Kozakova M, Kato K, Fraser AG. Arterial wave intensity and ventricular-arterial coupling by vascular ultrasound: rationale and methods for the automated analysis of forwards and backwards running waves. Ultrasound Med Biol. 2009 Feb;35(2):266-77. doi: 10.1016/j.ultrasmedbio.2008.08.013. Epub 2008 Nov 7. PMID 18992987
- [Background] Strauch AR, Berman MD, Miller HR. Substrate-associated macromolecules promote cytodifferentiation of BC3H1 myogenic cells. J Cell Physiol. 1991 Mar;146(3):337-48. doi: 10.1002/jcp.1041460302. PMID 1708777
- [Background] Ohte N, Saeki T, Miyabe H, Sakata S, Mukai S, Hayano J, Niki K, Sugawara M, Kimura G. Relationship between blood pressure obtained from the upper arm with a cuff-type sphygmomanometer and central blood pressure measured with a catheter-tipped micromanometer. Heart Vessels. 2007 Nov;22(6):410-5. doi: 10.1007/s00380-007-0998-5. Epub 2007 Nov 26. PMID 18044000
- [Background] Heart rate variability: standards of measurement, physiological interpretation and clinical use. Task Force of the European Society of Cardiology and the North American Society of Pacing and Electrophysiology. Circulation. 1996 Mar 1;93(5):1043-65. No abstract available. PMID 8598068
- [Background] Conraads VM, Pattyn N, De Maeyer C, Beckers PJ, Coeckelberghs E, Cornelissen VA, Denollet J, Frederix G, Goetschalckx K, Hoymans VY, Possemiers N, Schepers D, Shivalkar B, Voigt JU, Van Craenenbroeck EM, Vanhees L. Aerobic interval training and continuous training equally improve aerobic exercise capacity in patients with coronary artery disease: the SAINTEX-CAD study. Int J Cardiol. 2015 Jan 20;179:203-10. doi: 10.1016/j.ijcard.2014.10.155. Epub 2014 Oct 25. PMID 25464446
- [Background] Pinto R, Melo X, Angarten V, Pires ML, Borges M, Santos V, Abreu A, Santa-Clara H. The effects of 12-months supervised periodized training on health-related physical fitness in coronary artery disease: a randomized controlled trial. J Sports Sci. 2021 Aug;39(16):1893-1902. doi: 10.1080/02640414.2021.1907062. Epub 2021 Mar 28. PMID 33775203
- [Background] Kiviniemi AM, Hautala AJ, Kinnunen H, Tulppo MP. Endurance training guided individually by daily heart rate variability measurements. Eur J Appl Physiol. 2007 Dec;101(6):743-51. doi: 10.1007/s00421-007-0552-2. Epub 2007 Sep 12. PMID 17849143
- [Background] Vesterinen V, Nummela A, Heikura I, Laine T, Hynynen E, Botella J, Hakkinen K. Individual Endurance Training Prescription with Heart Rate Variability. Med Sci Sports Exerc. 2016 Jul;48(7):1347-54. doi: 10.1249/MSS.0000000000000910. PMID 26909534
- [Background] Manresa-Rocamora A, Sarabia JM, Javaloyes A, Flatt AA, Moya-Ramon M. Heart Rate Variability-Guided Training for Enhancing Cardiac-Vagal Modulation, Aerobic Fitness, and Endurance Performance: A Methodological Systematic Review with Meta-Analysis. Int J Environ Res Public Health. 2021 Sep 29;18(19):10299. doi: 10.3390/ijerph181910299. PMID 34639599
- [Background] Kavanagh T, Mertens DJ, Hamm LF, Beyene J, Kennedy J, Corey P, Shephard RJ. Prediction of long-term prognosis in 12 169 men referred for cardiac rehabilitation. Circulation. 2002 Aug 6;106(6):666-71. doi: 10.1161/01.cir.0000024413.15949.ed. PMID 12163425
- [Background] Kavanagh T, Mertens DJ, Hamm LF, Beyene J, Kennedy J, Corey P, Shephard RJ. Peak oxygen intake and cardiac mortality in women referred for cardiac rehabilitation. J Am Coll Cardiol. 2003 Dec 17;42(12):2139-43. doi: 10.1016/j.jacc.2003.07.028. PMID 14680741
- [Background] Witvrouwen I, Pattyn N, Gevaert AB, Possemiers N, Van Craenenbroeck AH, Cornelissen VA, Beckers PJ, Vanhees L, Van Craenenbroeck EM. Predictors of response to exercise training in patients with coronary artery disease - a subanalysis of the SAINTEX-CAD study. Eur J Prev Cardiol. 2019 Jul;26(11):1158-1163. doi: 10.1177/2047487319828478. Epub 2019 Feb 12. PMID 30755016
- [Background] Cornish AK, Broadbent S, Cheema BS. Interval training for patients with coronary artery disease: a systematic review. Eur J Appl Physiol. 2011 Apr;111(4):579-89. doi: 10.1007/s00421-010-1682-5. Epub 2010 Oct 23. PMID 20972578
- [Background] Villelabeitia-Jaureguizar K, Vicente-Campos D, Senen AB, Jimenez VH, Garrido-Lestache MEB, Chicharro JL. Effects of high-intensity interval versus continuous exercise training on post-exercise heart rate recovery in coronary heart-disease patients. Int J Cardiol. 2017 Oct 1;244:17-23. doi: 10.1016/j.ijcard.2017.06.067. Epub 2017 Jun 17. PMID 28648356
- [Background] Piepoli MF, Hoes AW, Agewall S, Albus C, Brotons C, Catapano AL, Cooney MT, Corra U, Cosyns B, Deaton C, Graham I, Hall MS, Hobbs FDR, Lochen ML, Lollgen H, Marques-Vidal P, Perk J, Prescott E, Redon J, Richter DJ, Sattar N, Smulders Y, Tiberi M, van der Worp HB, van Dis I, Verschuren WMM, Binno S; ESC Scientific Document Group. 2016 European Guidelines on cardiovascular disease prevention in clinical practice: The Sixth Joint Task Force of the European Society of Cardiology and Other Societies on Cardiovascular Disease Prevention in Clinical Practice (constituted by representatives of 10 societies and by invited experts)Developed with the special contribution of the European Association for Cardiovascular Prevention & Rehabilitation (EACPR). Eur Heart J. 2016 Aug 1;37(29):2315-2381. doi: 10.1093/eurheartj/ehw106. Epub 2016 May 23. No abstract available. PMID 27222591
- [Background] Vanhees L, Rauch B, Piepoli M, van Buuren F, Takken T, Borjesson M, Bjarnason-Wehrens B, Doherty P, Dugmore D, Halle M; Writing Group, EACPR. Importance of characteristics and modalities of physical activity and exercise in the management of cardiovascular health in individuals with cardiovascular disease (Part III). Eur J Prev Cardiol. 2012 Dec;19(6):1333-56. doi: 10.1177/2047487312437063. PMID 22637740
- [Background] Taylor JL, Bonikowske AR, Olson TP. Optimizing Outcomes in Cardiac Rehabilitation: The Importance of Exercise Intensity. Front Cardiovasc Med. 2021 Sep 3;8:734278. doi: 10.3389/fcvm.2021.734278. eCollection 2021. PMID 34540924
- [Background] Rauch B, Davos CH, Doherty P, Saure D, Metzendorf MI, Salzwedel A, Voller H, Jensen K, Schmid JP; 'Cardiac Rehabilitation Section', European Association of Preventive Cardiology (EAPC), in cooperation with the Institute of Medical Biometry and Informatics (IMBI), Department of Medical Biometry, University of Heidelberg, and the Cochrane Metabolic and Endocrine Disorders Group, Institute of General Practice, Heinrich-Heine University, Dusseldorf, Germany. The prognostic effect of cardiac rehabilitation in the era of acute revascularisation and statin therapy: A systematic review and meta-analysis of randomized and non-randomized studies - The Cardiac Rehabilitation Outcome Study (CROS). Eur J Prev Cardiol. 2016 Dec;23(18):1914-1939. doi: 10.1177/2047487316671181. Epub 2016 Oct 25. PMID 27777324
- [Background] Salzwedel A, Jensen K, Rauch B, Doherty P, Metzendorf MI, Hackbusch M, Voller H, Schmid JP, Davos CH. Effectiveness of comprehensive cardiac rehabilitation in coronary artery disease patients treated according to contemporary evidence based medicine: Update of the Cardiac Rehabilitation Outcome Study (CROS-II). Eur J Prev Cardiol. 2020 Nov;27(16):1756-1774. doi: 10.1177/2047487320905719. Epub 2020 Feb 23. PMID 32089005
- [Background] Winzer EB, Woitek F, Linke A. Physical Activity in the Prevention and Treatment of Coronary Artery Disease. J Am Heart Assoc. 2018 Feb 8;7(4):e007725. doi: 10.1161/JAHA.117.007725. No abstract available. PMID 29437600
- [Background] Badrov MB, Wood KN, Lalande S, Sawicki CP, Borrell LJ, Barron CC, Vording JL, Fleischhauer A, Suskin N, McGowan CL, Shoemaker JK. Effects of 6 Months of Exercise-Based Cardiac Rehabilitation on Autonomic Function and Neuro-Cardiovascular Stress Reactivity in Coronary Artery Disease Patients. J Am Heart Assoc. 2019 Sep 3;8(17):e012257. doi: 10.1161/JAHA.119.012257. Epub 2019 Aug 23. PMID 31438760
- [Background] Adams V, Reich B, Uhlemann M, Niebauer J. Molecular effects of exercise training in patients with cardiovascular disease: focus on skeletal muscle, endothelium, and myocardium. Am J Physiol Heart Circ Physiol. 2017 Jul 1;313(1):H72-H88. doi: 10.1152/ajpheart.00470.2016. Epub 2017 May 5. PMID 28476924
- [Background] Kotecha D, New G, Flather MD, Eccleston D, Pepper J, Krum H. Five-minute heart rate variability can predict obstructive angiographic coronary disease. Heart. 2012 Mar;98(5):395-401. doi: 10.1136/heartjnl-2011-300033. Epub 2011 Nov 25. PMID 22121069
- [Background] Huikuri HV, Stein PK. Heart rate variability in risk stratification of cardiac patients. Prog Cardiovasc Dis. 2013 Sep-Oct;56(2):153-9. doi: 10.1016/j.pcad.2013.07.003. Epub 2013 Aug 12. PMID 24215747
- [Background] Chen Y, Yu Y, Zou W, Zhang M, Wang Y, Gu Y. Association between cardiac autonomic nervous dysfunction and the severity of coronary lesions in patients with stable coronary artery disease. J Int Med Res. 2018 Sep;46(9):3729-3740. doi: 10.1177/0300060518778416. Epub 2018 Jun 25. PMID 29936852
- [Background] Adams V, Linke A, Krankel N, Erbs S, Gielen S, Mobius-Winkler S, Gummert JF, Mohr FW, Schuler G, Hambrecht R. Impact of regular physical activity on the NAD(P)H oxidase and angiotensin receptor system in patients with coronary artery disease. Circulation. 2005 Feb 8;111(5):555-62. doi: 10.1161/01.CIR.0000154560.88933.7E. PMID 15699275